CLINICAL TRIAL: NCT04681157
Title: Retrospective Study on Anosmias and Ageusias Linked to Infection by SARS-Cov 2
Brief Title: Retrospective Study on Anosmias and Ageusias Linked to Infection by Covid-19
Acronym: STras-Cov-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7754
Record Dates: First submitted 2020-12-22; First posted 2020-12-23 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Covid-19
Keywords: Covid-19; Odor disturbance; Taste disturbances; SARS-Cov2; Anosmia; Ageusia
MeSH Terms: conditions — COVID-19; Dysgeusia; Anosmia; Ageusia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Odor and taste disturbances have increased dramatically during this time of the COVID-19 pandemic. Currently, we have very little information on the demographic and clinical characteristics of the affected population, on the severity and course of the olfactory / taste loss.

The main objective of this research is to analyze the epidemiological, demographic and clinical characteristics of patients suspected or already confirmed of infection with SARS-Cov2 presenting with anosmia and / or ageusia.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Subject having had a loss of smell and / or taste that occurred during the period of the Covid-19 epidemic with or without other symptom (s) suggestive of a Covid infection -19
* Subject with suspected or confirmed Covid-19 infection
* Subject taken care of by the ENT service
* Subject not having expressed his opposition, after information, to the reuse of his data for the purposes of this research.

Exclusion Criteria:

* Subject having expressed opposition to participating in the study
* Subject under guardianship or guardianship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient having had a loss of smell and / or taste that occurred during the period of the Covid-19 epidemic with or without other symptom (s) suggestive of a Covid infection -19
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-03 (Actual); Primary Completion 2021-04-03 (Estimated); Study Completion 2021-04-03 (Estimated)

PRIMARY OUTCOMES:
Retrospective analysis of demographic and clinical characteristics of patients with suspected or already confirmed SARS-Cov2 infection with anosmia and / or ageusia | The files analysed retrospectily from February 01, 2020 to June 03, 2020 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Strasbourg University Hospitals - Otorhino-Laryngology Department, Strasbourg, Starsbourg, France